CLINICAL TRIAL: NCT02781532
Title: Evaluation of Predictive Visual Analog Scale (VAS) for Determining the Ingesta of Patients Carrying a Digestive Cancer
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 14-PP-05
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Digestive System Neoplasms
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of our study is to determine if the evaluation of ingesta of cancer patients by VAS (on the day of hospitalization) is able to predict the actual ingesta of patients during hospitalization (for patients malnourished, at risk of malnutrition or risk free).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Admitted to hospital for systemic therapy of gastrointestinal cancer
* Signature of the non-opposition.

Exclusion Criteria:

* Patients who because of their affection will fasted more than 12:00 during the three days preceding hospitalization.
* Artificial nutrition Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study has been proposed to all patients with a gastrointestinal cancer hospitalized in our service.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of ingesta | 3 days
  Evaluation of ingesta will be done using SAV scale.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, France, France

IPD SHARING:
Plan to Share IPD: No